CLINICAL TRIAL: NCT02236221
Title: Mechanism of Vitamin D in Influencing Offspring Obesity During Pregnancy
Brief Title: Effect of Vitamin D on Offspring Obesity
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xirong Guo, Vice-president of Nanjing Maternity and Child Health Care Hospital, Nanjing Medical University
Other Study IDs: NMU-530604-XG2
Record Dates: First submitted 2014-09-02; First posted 2014-09-10 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to observe the effect of lack or excess of Vitamin D in the first, second and third trimester on child birth weight, fat content and the secretion of metabolism related hormone, and clinical follow-up their offspring obesity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy women
* children
* Chinese

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with the early, mid and late pregnancy; Chilren
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
The level of Vitamin D of pregnancy women at second trimester | 20-24 weeks of pregnancy

SECONDARY OUTCOMES:
The level of Vitamin D of pregnancy women at first trimester | 12 weeks of pregnancy
The level of Vitamin D of pregnancy women at third trimester | 28-40 weeks of pregnancy
The birth weight, fat content and metabolism related hormone secretion of their offspring | At birth
The weight, fat content and metabolism related hormone secretion of their offspring at one year old | One years old
The weight, fat content and metabolism related hormone secretion of their offspring at 3 years old | 3 years old
The weight, fat content and metabolism related hormone secretion of their offspring at 5-7 years old | 5-7 years old
The weight, fat content and the secretion of metabolism related hormone of offspring at 18 years old | 18 years old

CONTACTS AND LOCATIONS:
Overall Officials: Xirong Guo, Dr., Principal Investigator — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu, China